CLINICAL TRIAL: NCT06253390
Title: Effect of the Metacognitive Training Programme (D-MCT) in Patients With Peripartum Depression
Brief Title: New Cognitive Treatment for Peripartum Depression
Acronym: MCT-DPP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PO23063*
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Postnatal Depression
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- D-MCT group (Active Comparator)
  Interventions: Behavioral: Metacognitive training
- DPN group (Other)
  Interventions: Behavioral: control

INTERVENTIONS:
Behavioral: Metacognitive training — Metacognitive training therapy
  Arms: D-MCT group
Behavioral: control — management technique as usual
  Arms: DPN group

SUMMARY:
The peripartum period is the period between the last month of pregnancy and up to a year after childbirth. It can be considered a difficult time for women, as it is a period of transition during which vulnerability to psychiatric disorders and in particular to major depressive disorder (MDD) (Vesga-Lopez, Blanco, Olfson, Grant & Hasin, 2008). Depression with peripartum onset (PPD) is characterised by the fact that the onset of symptoms may occur during pregnancy or within four weeks of delivery, but may also persist for up to 12 months after delivery (American Psychiatric Association, 2013). PPD affects 10 to 20% of women who have given birth (Tebeka et al. 2021). In addition, the psychological distress experienced by the mother during the peripartum period can disrupt interactions with her newborn (Lefkovics et al. 2014). Depression during this period can therefore have long-term consequences, not only for the women who suffer it, but also for their children (Gavin et al. 2005).

The investigators now know that women with PPD have deficits in metacognition. Metacognition is the body of knowledge, processes and practices that enable individuals to control and evaluate their own cognitive activities, thereby enabling them to regulate them (Flavell, 1976). Patients with PPD therefore have difficulty identifying, controlling and evaluating their own cognitive activities. These deficits may also represent a risk factor for the development of PPD if they are present at an early stage (Diop et al. 2022).

In patients with PPD, metacognitive therapies appear to be effective in reducing symptoms. In 2013, Bevan, Wittkowski and Wells conducted a pilot study to test the effects associated with metacognitive therapy in depression. This was the first published study to evaluate the effects of metacognitive therapy on patients with depression in the peripartum period. It shows promising results which it would be interesting to replicate, as this is a pilot study. A metacognitive training program for depression (D-MCT) was developed by Jelinek, Hauschildt, Moritz and Dubreucq in 2016, it is a brief group intervention that is easy to manage to participants. To date, no study has yet tested this specific program in patients with PPD, but it has been able to show its effectiveness in reducing the metacognitive deficits.

In the light of the scientific literature, the aims of this study are, firstly, to demonstrate the efficacy of D-MCT therapy in subjects with post-partum depression. Secondly, to examine the effects of this therapy on mother-child interactions.

The investigators make the following assumptions:

* Women in the experimental group showed a greater reduction in depressive symptoms and an improvement in metacognitive functioning than those in the control group.
* Women in the experimental group showed a reduction in depressive symptoms after therapy (v2) and maintenance of this improvement (v3).
* Improvement in the quality of mother-child bonding for women who took part in the program compared with those in the control group.
* Improvement in the quality of mother-child bonding after the program (v2 and v3) for women in the experimental group compared with when they entered the program.

DETAILED DESCRIPTION:
In peripartum depression (PPD), metacognition is affected, resulting in altered memories of parental experiences. The psychological distress endured by the mother during the peripartum period can disrupt interactions with her newborn. Depression during this period can have long-term consequences, not only for the women who suffers it, but also for their children (3). In an attempt to prevent the deleterious consequences of PPD, a number of treatment techniques have been shown to be effective. These include not only antidepressants, but also psychological supports. Cognitive behavioural therapy (CBT) was shown in a meta-analysis to be significantly associated with a reduction in symptoms on the Edinburgh Postnatal Depression Scale. However, although this meta-analysis showed a reduction in depressive symptoms, it did not demonstrate a significant reduction in anxiety symptoms specific to PPD. Most of the studies carried out to date on the efficacy of CBT in the treatment of PPD focus essentially on depressive symptoms, which could explain the relapse after six months. In order to minimise the risk of relapse, it would be worthwhile turning to a therapy that is effective on both depressive and anxiety symptoms. One therapy that could be adapted to this type of care is metacognitive therapy (MCT). Normann, Emmerik and Morina in 2014 showed the effectiveness of metacognitive therapy on anxiety and depression through their meta-analysis. The meta-analysis included 384 patients suffering from anxiety and depression. This study showed that MCT was effective in the treatment of both anxiety disorders and depression. The study also showed that MCT was more effective than cognitive behavioural therapy. The authors also demonstrated that maladaptive metacognitive beliefs were responsible for maintaining psychological distress. In other words, acting on maladaptive metacognitive processes would enable MCT to be effective. In patients with PPD, metacognitive therapies also appear to be effective in reducing symptoms. Bevan, Wittkowski and Wells in 2013 carried out a pilot study to test the effects associated with this metacognitive therapy in peripartum depression. The results showed a significant reduction in symptoms of anxiety and depression. This pilot study provides preliminary evidence that metacognitive therapy is associated with significant improvements in PPD symptoms. The results of this pilot study are promising and call for a case-control study with a larger sample of patients and a form of metacognitive therapy developed specifically for the management of PDD (Metacognitive Training Therapy, D-MCT) by Stephen Moritz's team (University Medical Center Hamburg-Eppendorf, Department of Psychiatry and Psychotherapy, Hamburg, Germany) and translated into French by Julien Dubreucq (Centre Référent de Réhabilitation Psychosociale et de Remédiation Cognitive (C3R), Centre Hospitalier Alpes Isère, Grenoble).

D-MCT is a brief group intervention that is easy to manage to participants. The program proved to be well accepted by participants, with high acceptance rates. The program not only proved feasible and acceptable, but also effective in reducing cognitive biases and rumination and increasing self-esteem.

In view of the efficacy of this programme in patients presenting with a characterised depressive episode, it seems essential to test it in patients with PPD by comparing it in a prospective randomised study with a non-metacognitive group usually practised in the department (control group). Our main objective is therefore to find out, without any preconceived ideas, whether D-MCT therapy is more effective than the usual treatment (control group) in reducing depressive symptoms during the peripartum period. The secondary objective is to determine the impact of D-MCT on the attachment relationship between mother and child.

ELIGIBILITY:
Inclusion Criteria:

* Women over 18 years
* Meets the diagnostic criteria for depressive disorder with peripartum onset (PPD) (APA, 2013) and has already given birth
* EPDS score over 10
* Have given their consent to take part in the study
* Be affiliated to a social security system
* Have an adequate knowledge of written, understood and spoken French (French mother tongue or primary education in the French education system) All women with PPD, whether breastfeeding or not, can be included in the study. Baby care can be organised if mothers are unable to have their babies looked after. This service is provided by nurses from the UPPE in the unit's reception room, which has all the equipment needed to care for infants. Mothers meet the nurses before the group and tell them what they expect, and the nurses give them feedback when they come to collect their baby.

Exclusion Criteria:

* - Be the subject of a protection measure
* Being a minor
* Meets the diagnostic criteria for schizophrenia spectrum disorders (brief psychotic disorder; schizophrenic disorder; schizoaffective disorder; delusional disorder; brief psychotic disorder with peripartum onset)
* Meet the criteria for substance abuse or dependence (alcohol, drugs)
* With insufficient command of the French language
* People with a deceased child
* People who do not meet the diagnostic criteria for depressive disorder with peripartum onset (APA, 2013)
* People who do not agree to take part in the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Edinburgh Postnatal Depression Scale score | 3 months
  Edinburgh Postnatal Depression Scale (EPDS), Cox, Holdent & Sagovsky, 1987, translated and validated in French by Guedeney & Fermanian, 1998.
  the minimum value is 0 and maximum value is 30. Higher scores mean a worse outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

IPD SHARING:
Plan to Share IPD: No